CLINICAL TRIAL: NCT02619396
Title: Radiofrequency Power, Lesion Size Index and Oesophageal Temperature Alerts During Atrial Fibrillation Ablation: A Pilot Study
Brief Title: RF Power, LSI and Oesophageal Temperature Alerts During AF Ablation (PiLOT-AF Study)
Acronym: PiLOT-AF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oxford University Hospitals NHS Trust (Other)
Responsible Party: Principal Investigator, Dr Tim Betts MD MBChB FRCP, Consultant Cardiologist and Electrophysiologist, Oxford University Hospitals NHS Trust
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11536-SPON
Record Dates: First submitted 2015-10-26; First posted 2015-12-02 (Estimated); Results first posted 2020-07-08 (Actual); Last update posted 2020-07-08 (Actual); Status verified 2020-07

CONDITIONS: Atrial Fibrillation
Keywords: radiofrequency power; lesion size index; esophageal temperature alerts
MeSH Terms: conditions — Atrial Fibrillation | interventions — Laser Speckle Contrast Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group "20 W / LSI 4" (Active Comparator): Patients elected to atrial fibrillation (AF) ablation and randomized to Combination 1 of radiofrequency (RF) power and Lesion Size Index (LSI) on left atrial (LA) posterior wall
  Interventions: Procedure: Combination 1 of radiofrequency (RF) power and Lesion Size Index (LSI) on left atrial (LA) posterior wall
- Group "40 W / LSI 4" (Active Comparator): Patients elected to atrial fibrillation (AF) ablation and randomized to Combination 2 of radiofrequency (RF) power and Lesion Size Index (LSI) on left atrial (LA) posterior wall
  Interventions: Procedure: Combination 2 of radiofrequency (RF) power and Lesion Size Index (LSI) on left atrial (LA) posterior wall
- Group "20 W / LSI 5" (Active Comparator): Patients elected to atrial fibrillation (AF) ablation and randomized to Combination 3 of radiofrequency (RF) power and Lesion Size Index (LSI) on left atrial (LA) posterior wall
  Interventions: Procedure: Combination 3 of radiofrequency (RF) power and Lesion Size Index (LSI) on left atrial (LA) posterior wall
- Group "40 W / LSI 5" (Active Comparator): Patients elected to atrial fibrillation (AF) ablation and randomized to Combination 4 of radiofrequency (RF) power and Lesion Size Index (LSI) on left atrial (LA) posterior wall
  Interventions: Procedure: Combination 4 of radiofrequency (RF) power and Lesion Size Index (LSI) on left atrial (LA) posterior wall

INTERVENTIONS:
Procedure: Combination 1 of radiofrequency (RF) power and Lesion Size Index (LSI) on left atrial (LA) posterior wall — 20 W RF power and target LSI = 4 on LA posterior wall
  Arms: Group "20 W / LSI 4"
Procedure: Combination 2 of radiofrequency (RF) power and Lesion Size Index (LSI) on left atrial (LA) posterior wall — 40 W RF power and target LSI = 4 on LA posterior wall
  Arms: Group "40 W / LSI 4"
Procedure: Combination 3 of radiofrequency (RF) power and Lesion Size Index (LSI) on left atrial (LA) posterior wall — 20 W RF power and target LSI = 5 on LA posterior wall
  Arms: Group "20 W / LSI 5"
Procedure: Combination 4 of radiofrequency (RF) power and Lesion Size Index (LSI) on left atrial (LA) posterior wall — 40 W RF power and target LSI = 5 on LA posterior wall
  Arms: Group "40 W / LSI 5"

SUMMARY:
Atrial fibrillation (AF) is a very common abnormal heart rhythm, triggered by rapid electrical activity originating from the pulmonary veins (PVs) that drain blood from the lungs back to the left atrium (LA). Ablation of the junction between the PVs and the LA, electrically isolating the veins from the heart, is the key to prevent AF.

When using radiofrequency energy (RF), transmural lesions are required to achieve permanent pulmonary vein isolation (PVI). New technologies are currently available to predict the ablation lesion depth and to guide the duration of each application. However, deeper lesions mean a higher risk of overheating and damage of adjacent structures such as the esophagus that lies against the back wall of the LA. In order to minimize this risk, the investigators continuously monitor the temperature inside the esophagus during the procedure through a probe placed in the esophagus and they promptly terminate energy delivery in case of any esophageal temperature rises more than 39°C.

To date, it is not known if a low power for a longer time is better than a high power for a shorter time when ablating on the LA posterior wall in order to create permanent scars without heating the esophagus.

Therefore, the investigators plan to compare the incidence of esophageal temperature alerts and the success of the procedure with four different energy settings during ablation on the LA posterior wall.

DETAILED DESCRIPTION:
The PiLOT-AF study is a prospective single-centre randomized observational study aiming at comparing different radiofrequency energy (RF) settings during atrial fibrillation (AF) ablation on the left atrial (LA) posterior wall, in terms of esophageal heating, acute and long-term procedure success and procedural complications.

Patients scheduled for their first RF ablation, because of a history of symptomatic and drug-refractory paroxysmal or persistent AF, will be considered for inclusion in the study.

Potential subjects will initially be approached 4-6 weeks before their ablation procedure, in order to give them enough time to consider the information, to ask questions to the investigators, their family doctor or other independent parties to decide whether they wish to participate in the study or not.

For those interested in participation, a baseline assessment will be arranged to coincide with their standard pre-admission visit, for informed consent, screening and eligibility assessment and randomization.

All AF ablation procedures will be performed in a standard fashion, under general anaesthesia and with continuous esophageal temperature monitoring using a sinusoidal multi-sensor esophageal temperature probe (CIRCAtemp). After LA geometry reconstruction using 3-dimensional electroanatomical mapping EnSite Velocity and a multipolar circular mapping catheter St Jude Medical Optima, the ablation catheter Endosense Tacticath through a deflectable sheath St Medical Agilis will be used for Pulmonary Vein Isolation (PVI). Standardized RF settings will be used during ablation on the LA anterior wall as current practice in our centre. Different RF settings will be used on the LA posterior wall, according to randomization group. Moreover target values will be chosen for Lesion Size Index (LSI), a parameter useful to predict the lesion depth, during ablation on LA posterior wall. The duration of RF delivery on the LA posterior wall will be dictated by achievement of the target LSI or esophageal temperature rise > 39◦C during ablation. PVI will be achieved and confirmed after 30 minutes waiting time. In case of acute PV reconnection, ablation at sites of breakthrough signals will be performed in order to achieve durable PVI. The occurrence of acute PV reconnection (PVR) with sites of breakthrough signals on the LA posterior wall will be recorded for each procedure. The total procedure and RF ablation times will be also collected.

After the ablation, before discharge the symptoms status and heart rhythm will be assessed and the patient will be instructed to commence a symptoms diary. Telephone follow-ups will be then performed at 3 and 6 months to assess current symptom status. Standard care follow-up Arrhythmia Clinic visits will be also performed 3-4 months after the ablation procedure. Ad hoc visits and/or additional investigations as prolonged electrocardiogram (ECG) monitoring will also take place, dictated by arrhythmia symptoms and assessment for potential adverse events related to the procedure, in accordance with standard practice.

The end of the study for each patient will be the date of the 6 months telephone follow-up.

ELIGIBILITY:
Inclusion Criteria:

* male or female, aged 18 to 80 years;
* willing and able to give informed consent for participation in the study;
* history of symptomatic and drug-refractory atrial fibrillation;
* planned atrial fibrillation (AF) ablation on a clinical basis.

Exclusion Criteria:

* previous AF ablation;
* pregnancy, trying for a baby or breast feeding;
* oesophageal obstruction (mass, stricture), diverticulum or varices, tracheo-oesophageal fistula or any other oesophageal conditions prohibiting the use of oesophageal temperature probe for continuous luminal temperature monitoring;
* any other significant disease or disorder which, in the opinion of the investigator, may either put the participants at risk because of participation in the study, or may influence the result of the study, or the participant's ability to participate in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2016-01; Primary Completion 2017-03-11 (Actual); Study Completion 2017-03-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tim R Betts, MD, Principal Investigator — Oxford University Hospitals NHS Trust
Locations (1):
- John Radcliffe Hospital, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Petersen HH, Chen X, Pietersen A, Svendsen JH, Haunso S. Tissue temperatures and lesion size during irrigated tip catheter radiofrequency ablation: an in vitro comparison of temperature-controlled irrigated tip ablation, power-controlled irrigated tip ablation, and standard temperature-controlled ablation. Pacing Clin Electrophysiol. 2000 Jan;23(1):8-17. doi: 10.1111/j.1540-8159.2000.tb00644.x. PMID 10666748
- [Background] Haines DE. Determinants of lesion size during radiofrequency catheter ablation: the role of electrode-tissue contact pressure and duration of energy delivery. Journal of Cardiovascular Electrophysiology. 2008;2(6):509-15.
- [Background] Kautzner J, Neuzil P, Peickl P. Contact force, FTI and Lesion continuity are critical to improve durable PV isolation: EFFICAS 2 results. Heart Rhythm. 2012;9(5S):1-564
- [Background] Cummings JE, Schweikert RA, Saliba WI, Burkhardt JD, Brachmann J, Gunther J, Schibgilla V, Verma A, Dery M, Drago JL, Kilicaslan F, Natale A. Assessment of temperature, proximity, and course of the esophagus during radiofrequency ablation within the left atrium. Circulation. 2005 Jul 26;112(4):459-64. doi: 10.1161/CIRCULATIONAHA.104.509612. Epub 2005 Jul 18. PMID 16027254
- [Background] Singh SM, d'Avila A, Doshi SK, Brugge WR, Bedford RA, Mela T, Ruskin JN, Reddy VY. Esophageal injury and temperature monitoring during atrial fibrillation ablation. Circ Arrhythm Electrophysiol. 2008 Aug;1(3):162-8. doi: 10.1161/CIRCEP.107.789552. PMID 19808410
- [Background] Kowalski M, Grimes MM, Perez FJ, Kenigsberg DN, Koneru J, Kasirajan V, Wood MA, Ellenbogen KA. Histopathologic characterization of chronic radiofrequency ablation lesions for pulmonary vein isolation. J Am Coll Cardiol. 2012 Mar 6;59(10):930-8. doi: 10.1016/j.jacc.2011.09.076. PMID 22381429
- [Derived] Leo M, Pedersen M, Rajappan K, Ginks MR, Hunter RJ, Bowers R, Kalla M, Bashir Y, Betts TR. Power, Lesion Size Index and Oesophageal Temperature Alerts During Atrial Fibrillation Ablation: A Randomized Study. Circ Arrhythm Electrophysiol. 2020 Oct;13(10):e008316. doi: 10.1161/CIRCEP.120.008316. Epub 2020 Sep 8. PMID 32898435

RESULTS

PARTICIPANT FLOW:
Groups:
- Group "20 W / LSI 4": Patients elected to AF ablation and randomized to Combination 1 of RF power and LSI on LA posterior wall
  Combination 1 of RF power and LSI on LA posterior wall: 20 W RF power and target LSI = 4 on LA posterior wall
- Group "40 W / LSI 4": Patients elected to AF ablation and randomized to Combination 2 of RF power and LSI on LA posterior wall
  Combination 2 of RF power and LSI on LA posterior wall: 40 W RF power and target LSI = 4 on LA posterior wall
- Group "20 W / LSI 5": Patients elected to AF ablation and randomized to Combination 3 of RF power and LSI on LA posterior wall
  Combination 3 of RF power and LSI on LA posterior wall: 20 W RF power and target LSI = 5 on LA posterior wall
- Group "40 W / LSI 5": Patients elected to AF ablation and randomized to Combination 4 of RF power and LSI on LA posterior wall
  Combination 4 of RF power and LSI on LA posterior wall: 40 W RF power and target LSI = 5 on LA posterior wall
Period: Overall Study
Arm/Group | Group "20 W / LSI 4" | Group "40 W / LSI 4" | Group "20 W / LSI 5" | Group "40 W / LSI 5"
Started | 20 | 20 | 20 | 20
Completed | 20 | 20 | 20 | 20
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Group "20 W / LSI 4": Patients elected to AF ablation and randomized to Combination 1 of RF power and Lesion Size Index (LSI) on LA posterior wall: 20 W RF power and target LSI = 4 on LA posterior wall
- Group "40 W / LSI 4": Patients elected to AF ablation and randomized to Combination 2 of RF power and Lesion Size Index (LSI) on LA posterior wall: 40 W RF power and target LSI = 4 on LA posterior wall
- Group "20 W / LSI 5": Patients elected to AF ablation and randomized to Combination 3 of RF power and Lesion Size Index (LSI) on LA posterior wall: 20 W RF power and target LSI = 5 on LA posterior wall
- Group "40 W / LSI 5": Patients elected to AF ablation and randomized to Combination 4 of RF power and Lesion Size Index (LSI) on LA posterior wall: 40 W RF power and target LSI = 5 on LA posterior wall
- Total: Total of all reporting groups
Arm/Group | Group "20 W / LSI 4" | Group "40 W / LSI 4" | Group "20 W / LSI 5" | Group "40 W / LSI 5" | Total
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.9 (9.2) | 60.1 (9.4) | 55.7 (10) | 61.3 (9.6) | 59.0 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 8 | 6 | 6 | 21
  Male | 19 | 12 | 14 | 14 | 59
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United Kingdom | 20 | 20 | 20 | 20 | 80
Paroxysmal atrial fibrillation (AF) [Count of Participants; unit: Participants] | 9 | 8 | 6 | 8 | 31
Atrial fibrillation (AF) history duration (months) [Median (Inter-Quartile Range); unit: months] | 24 [17 to 44] | 27 [18 to 48] | 20 [17 to 44] | 24 [21 to 45] | 24 [17 to 44]
Body Mass Index (BMI) [Mean (Standard Deviation); unit: BMI unit = kg/m^2] | 30.8 (4.6) | 27.3 (5) | 28.2 (4.85) | 28.8 (4.9) | 29.2 (6.3)
Left atrial (LA) size [Mean (Standard Deviation); unit: diameter (mm)] | 43 (6) | 41.4 (6.5) | 42.4 (7.7) | 43.7 (9.3) | 42.8 (7.4)
Left ventricular (LV) function [Mean (Standard Deviation); unit: LVEF (%)] | 60 (11.5) | 60 (9.2) | 60 (10.2) | 57.9 (6.4) | 59.4 (9.2)

OUTCOME MEASURES:

1. Primary Outcome: Rate of Oesophageal Temperature Alerts During Radiofrequency Energy (RF) Ablation on the Left Atrial (LA) Posterior Wall
Description: Number of patients with luminal oesophageal temperature rises > 39◦C during radiofrequency (RF) ablation on the left atrial (LA) posterior wall
Time Frame: 1 day
Measure: Count of Participants; unit: Participants
Groups:
- Group "20 W / LSI 4": Patients elected to atrial fibrillation (AF) ablation and randomized to Combination 1 of radiofrequency energy (RF) power and Lesion Size Index (LSI) on left atrial (LA) posterior wall
  Combination 1 of radiofrequency energy (RF) power and lesion Size Index (LSI) on LA posterior wall: 20 W RF power and target LSI = 4 on LA posterior wall
- Group "40 W / LSI 4": Patients elected to atrial fibrillation (AF) ablation and randomized to Combination 2 of radiofrequency energy (RF) power and Lesion Size Index (LSI) on left atrial (LA) posterior wall
  Combination 2 of radiofrequency energy (RF) power and lesion Size Index (LSI) on LA posterior wall: 40 W RF power and target LSI = 4 on LA posterior wall
- Group "20 W / LSI 5": Patients elected to atrial fibrillation (AF) ablation and randomized to Combination 3 of radiofrequency energy (RF) power and Lesion Size Index (LSI) on left atrial (LA) posterior wall
  Combination 3 of radiofrequency energy (RF) power and lesion Size Index (LSI) on LA posterior wall: 20 W RF power and target LSI = 5 on LA posterior wall
- Group "40 W / LSI 5": Patients elected to atrial fibrillation (AF) ablation and randomized to Combination 4 of radiofrequency energy (RF) power and Lesion Size Index (LSI) on left atrial (LA) posterior wall
  Combination 4 of radiofrequency energy (RF) power and lesion Size Index (LSI) on LA posterior wall: 40 W RF power and target LSI = 5 on LA posterior wall
Arm/Group | Group "20 W / LSI 4" | Group "40 W / LSI 4" | Group "20 W / LSI 5" | Group "40 W / LSI 5"
Number analyzed (Participants) | 20 | 20 | 20 | 20
Participants | 18 | 18 | 19 | 19

2. Primary Outcome: Oesophageal Temperature Alerts Per Patient
Description: Number of oesophageal temperature alerts per patient
Time Frame: 1 day
Measure: Median (Inter-Quartile Range); unit: oesophageal temperature alerts
Arm/Group | Group "20 W / LSI 4" | Group "40 W / LSI 4" | Group "20 W / LSI 5" | Group "40 W / LSI 5"
Number analyzed (Participants) | 20 | 20 | 20 | 20
oesophageal temperature alerts | 4 [2 to 8] | 4 [2 to 6] | 7 [5 to 10] | 4 [2 to 6]

3. Secondary Outcome: Rate of First-pass Pulmonary Vein Isolation (PVI)
Description: Rate of Pulmonary Veins (PVs) isolated after completion of first Pulmonary Vein Encirclement
Time Frame: 1 day
Population: 80 pulmonary veins in each group (4 veins per patient, 20 patients)
Measure: Number; unit: pulmonary veins
Units Other Than Participants: number of pulmonary veins in each group
Arm/Group | Group "20 W / LSI 4" | Group "40 W / LSI 4" | Group "20 W / LSI 5" | Group "40 W / LSI 5"
Number analyzed (Participants) | 20 | 20 | 20 | 20
Number analyzed (number of pulmonary veins in each group) | 80 | 80 | 80 | 80
pulmonary veins | 59 | 59 | 38 | 59

4. Secondary Outcome: Rate of Acute Pulmonary Vein Reconnection (PVR)
Description: Number of pulmonary veins acutely reconnected after catheter ablation and isolation
Time Frame: 1 day
Population: 80 pulmonary veins in each group (4 veins per patient, 20 patients)
Measure: Number; unit: pulmonary veins
Units Other Than Participants: number of pulmonary veins in each group
Groups:
- Group "20 W / LSI 5": Patients elected to atrial fibrillation (AF) ablation and randomized to Combination 3 of radiofrequency energy (RF) power and Lesion Size Index (LSI) on left atrial (LA) posterior wall
  Combination 3of radiofrequency energy (RF) power and lesion Size Index (LSI) on LA posterior wall: 20 W RF power and target LSI = 5 on LA posterior wall
Arm/Group | Group "20 W / LSI 4" | Group "40 W / LSI 4" | Group "20 W / LSI 5" | Group "40 W / LSI 5"
Number analyzed (Participants) | 20 | 20 | 20 | 20
Number analyzed (number of pulmonary veins in each group) | 80 | 80 | 80 | 80
pulmonary veins | 5 | 10 | 17 | 5

5. Secondary Outcome: Total Procedure Time
Description: Total duration of the procedure
Time Frame: 1 day
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Group "20 W / LSI 4" | Group "40 W / LSI 4" | Group "20 W / LSI 5" | Group "40 W / LSI 5"
Number analyzed (Participants) | 20 | 20 | 20 | 20
minutes | 180 [131.3 to 218] | 165 [145 to 180] | 180 [156.3 to 210] | 165 [146.3 to 191.3]

6. Secondary Outcome: Total Radiofrequency Energy (RF) Time for Pulmonary Vein Isolation (PVI)
Description: Total duration of radiofrequency energy required to achieve electrical isolation of the pulmonary veins
Time Frame: 1 day
Population: Patients/ablation procedures per group
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Group "20 W / LSI 4" | Group "40 W / LSI 4" | Group "20 W / LSI 5" | Group "40 W / LSI 5"
Number analyzed (Participants) | 20 | 20 | 20 | 20
minutes | 28.4 [25.2 to 40.1] | 23.8 [16.9 to 34.7] | 38 [28.4 to 46.3] | 22 [18.7 to 33.8]

7. Secondary Outcome: Freedom From Atrial Fibrillation
Description: Absence of symptoms suggestive of atrial fibrillation and no documentation of atrial fibrillation during the follow-up period
Time Frame: 6 months after the procedure
Population: Patients per group
Measure: Count of Participants; unit: Participants
Arm/Group | Group "20 W / LSI 4" | Group "40 W / LSI 4" | Group "20 W / LSI 5" | Group "40 W / LSI 5"
Number analyzed (Participants) | 20 | 20 | 20 | 20
Participants | 8 | 3 | 7 | 2

8. Secondary Outcome: Esophageal Symptoms After the Atrial Fibrillation (AF) Ablation
Description: Difficult or painful swallowing, heartburn, acid reflux, sore throat, hoarseness, cough, nausea, vomiting, non-cardiac chest pain
Time Frame: 6 months after the procedure
Population: Patients per group
Measure: Count of Participants; unit: Participants
Arm/Group | Group "20 W / LSI 4" | Group "40 W / LSI 4" | Group "20 W / LSI 5" | Group "40 W / LSI 5"
Number analyzed (Participants) | 20 | 20 | 20 | 20
Participants | 0 | 0 | 0 | 0

9. Other Pre Specified Outcome: Procedural Complications
Description: Pericardial effusion, transient ischemic attack/stroke, phrenic nerve injury, pulmonary vein stenosis, open-heart surgery, death
Time Frame: 1 day
Measure: Count of Participants; unit: Participants
Arm/Group | Group "20 W / LSI 4" | Group "40 W / LSI 4" | Group "20 W / LSI 5" | Group "40 W / LSI 5"
Number analyzed (Participants) | 20 | 20 | 20 | 20
Participants | 0 | 1 | 0 | 1

ADVERSE EVENTS:
Time Frame: 6 months
Description: Regular investigator assessment before discharge after catheter ablation and at subsequent telephone follow-ups
Arm/Group | Group "20 W / LSI 4" | Group "40 W / LSI 4" | Group "20 W / LSI 5" | Group "40 W / LSI 5"
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20 | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 1/20 | 0/20 | 1/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20 | 0/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group "20 W / LSI 4" (N=20) | Group "40 W / LSI 4" (N=20) | Group "20 W / LSI 5" (N=20) | Group "40 W / LSI 5" (N=20)
Stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-03-10): https://cdn.clinicaltrials.gov/large-docs/96/NCT02619396/Prot_SAP_000.pdf